CLINICAL TRIAL: NCT02893137
Title: Enhancing Optune Therapy of Recurrent Glioblastoma Multiforme Using Targeted Surgical Skull Remodeling
Brief Title: Enhancing Optune Therapy With Targeted Craniectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 54762
Record Dates: First submitted 2016-08-22; First posted 2016-09-08 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2016-08

CONDITIONS: Glioblastoma
Keywords: Tumour treating fields; Optune; Craniectomy; TTFields
MeSH Terms: conditions — Glioblastoma | interventions — Craniotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Craniectomy and Optune (Experimental): Patients will receive best physician's choice chemotherapy along with Optune therapy and craniotomy surgery. Optune therapy will be administered in the standard configuration and in accordance with current guidelines with the exception of the surgical intervention.
  Interventions: Device: Optune; Procedure: Craniectomy

INTERVENTIONS:
Device: Optune — For further information see www.optune.com
  Other Names: NovoTTF-100A; Tumor treating fields; TTFields
Procedure: Craniectomy — A small hole is placed in the skull between the tumor and the closest Optune electrode. The position and geometry of the craniotomy is determined by computersimulation of the electric field induced by Optune therapy. Craniotomy is a surgical procedure, which is carried out under general anaesthesia.

SUMMARY:
The present study proposes a new and potentially superior clinical approach to Optune™ therapy of selected glioblastoma patients. The approach is based on combining TTFields with targeted surgical skull remodeling, such as minor craniectomy or a distribution of burr holes, designed for the individual patient. Pre-clinical modeling results suggest that such procedures may enhance the induced electrical field strength by up to ~100% and thereby potentially improve the clinical outcome of treated patients to a significant extent.

The study is an open label phase 1 clinical pilot experiment designed to investigate feasibility, safety and efficacy of the concept. Fifteen patients with first recurrence of glioblastoma will be included in the trial. All patients will receive TTFields therapy with targeted craniotomy and best physician's choice chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathological evidence of GBM using WHO classification criteria
* Estimated survival minimum three months
* Supratentorial tumor
* Not a candidate for further radiotherapy
* First disease recurrence in accordance with RANO criteria
* Karnofsky scale score minimum 70
* Ability to comply with Optune therapy
* Tumor characteristics which indicate significant expected benefit from feasible craniotomy or skull remodelling surgery combined with TTFields
* Focal tumor
* Most superficial border of tumor or resection cavity closer than 2 cm from brain surface
* Use of validated anti-conception for female participants in accordance with guidelines provided by the Danish Health and Medicines Authority
* Signed written consent form

Exclusion Criteria:

* Pregnancy or nursing. Fertile female participants will be required to take a validated pregnancy test for evaluation of pregnancy
* Less than four weeks since radiation therapy
* Infratentorial tumor
* Implanted pacemaker, programmable shunt, defibrillator, deep brain stimulator, other implanted devices in the brain, or documented clinically significant arrhythmias.
* Uncontrollable symptomatic epilepsy, refractory to standard medication. Epilepsy will not necessarily contraindicate participation in the trial as this is a common complication to the disease. Eligibility will be determined by the examining physician and investigators in conjunction upon careful consideration of patient safety.
* Contraindications for skull remodelling surgery, e.g. bleeding diathesis or severe infection.
* Significant co-morbidities (within four weeks prior to enrolment)
* Significant liver function impairment - ALT > 3 times the upper limit of normal
* Total bilirubin > upper limit of normal
* Significant renal impairment (serum creatinine > 1.7 mg/dL)
* Coagulopathy (as evidenced by PT or APTT > 1.5 times control in normal individuals not undergoing anticoagulation)
* Thrombocytopenia (platelet count < 100x10^3/μL )
* Anemia (Hb < 10 g/L)
* Active participation in another clinical treatment trial

Patients will be regarded as participants when they have signed a consent form and have been found suitable for enrolment by the examining physician, in accordance with the abovecriteria. Patients may receive medication depending on their clinical condition and other diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Frequency of serious adverse events | Through study completion, an average of 18 months.
  Based on CTCAE.

SECONDARY OUTCOMES:
Overall survival | Through study completion, an average of 18 months.
Progression free survival | Through study completion, an average of 18 months.
Progression free survival at six months | Through study completion, an average of 18 months.
% 1-year survival | Through study completion, an average of 18 months.
Objective response rate | Will be assessed at baseline and upon clinical follow-up every 3rd month until exclusion. Data will be presented at trial termination.
  Assessed by RANO criteria
Quality of life | Will be assessed at baseline and upon clinical follow-up every 3rd month until exclusion. Data will be presented at trial termination.
  Assessed by EORTC QLQ-30 and QLQ-BN20
Cumulative corticosteroid dosage | Will be assessed at baseline and upon clinical follow-up every 3rd month until exclusion. Data will be presented at trial termination.
Karnofsky performance score | Will be assessed at baseline and upon clinical follow-up every 3rd month until exclusion. Data will be presented at trial termination.

CONTACTS AND LOCATIONS:
Overall Officials: Anders R Korshoej, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus C, Aarhus, Denmark

REFERENCES:
- [Derived] Korshoej AR, Sorensen JCH, von Oettingen G, Poulsen FR, Thielscher A. Optimization of tumor treating fields using singular value decomposition and minimization of field anisotropy. Phys Med Biol. 2019 Feb 8;64(4):04NT03. doi: 10.1088/1361-6560/aafe54. PMID 30641498